CLINICAL TRIAL: NCT04901624
Title: Use of Behavioral Economics in Repeat SARS-CoV-2 (COVID-19) Antibody Testing in Disadvantaged Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: AltaMed Health Services Corporation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-20-00793; 3R33AG057395-04S1 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-05-25 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: SARS-CoV-2
Keywords: antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Personal Risk + Loss Protection (Experimental): Personal Risk + Loss Protection
  Interventions: Behavioral: Personal Risk Messaging; Behavioral: Loss Protection
- Personal Risk + Lottery Incentive (Experimental): Personal Risk + Lottery Incentive
  Interventions: Behavioral: Personal Risk Messaging; Behavioral: Lottery Incentive
- Family Risk + Loss Protection (Experimental): Family Risk + Loss Protection
  Interventions: Behavioral: Family Risk Messaging; Behavioral: Loss Protection
- Family Risk + Lottery Incentive (Experimental): Family Risk + Lottery Incentive
  Interventions: Behavioral: Family Risk Messaging; Behavioral: Lottery Incentive

INTERVENTIONS:
Behavioral: Family Risk Messaging — Family risk framing may engender concern for loved ones. It may also make it easier to mentally simulate family burdens with COVID-19 such as knowing how several people in the family becoming sick could adversely affect the lives of everyone in the family. Households randomized to family risk messaging will receive the following message: "Antibody testing will help you understand your family's risk of getting COVID-19."
  Arms: Family Risk + Loss Protection; Family Risk + Lottery Incentive
Behavioral: Personal Risk Messaging — Personal risk framing may engender concern for oneself. Households randomized to personal risk messaging will receive the following message: "Antibody testing will help you understand your risk of getting COVID-19."
  Arms: Personal Risk + Loss Protection; Personal Risk + Lottery Incentive
Behavioral: Loss Protection — Household members are offered a baseline incentive with a 90% (9 in 10) chance of $60 and receive insurance on winning the baseline incentive for repeat antibody testing.
  Arms: Family Risk + Loss Protection; Personal Risk + Loss Protection
Behavioral: Lottery Incentive — Household members are offered a baseline incentive with a 90% (9 in 10) chance of $60 and receive a bonus lottery incentive with a 4 small (1 in 25) chance of winning $150 for repeat antibody testing.
  Arms: Family Risk + Lottery Incentive; Personal Risk + Lottery Incentive

SUMMARY:
Repeat testing for SARS-CoV-2 antibodies in disadvantaged communities will help identify active and recovered infections over time, and as more is understood about antibody protection, it may help identify persons who have immunity. Many questions about social barriers and behavioral facilitators remain unanswered. This project aims to evaluate the effectiveness of risk-based messaging and incentives that promote repeated testing for SARS-CoV-2 antibodies, as well as to understand social and behavioral determinants of COVID-19 testing and variations within sub-groups of this population.

DETAILED DESCRIPTION:
The rapid spread of the SARS-CoV-2 virus has greatly impacted underserved populations. This project aims to understand social and behavioral determinants of COVID-19 testing and variations within sub-groups of this population. In partnership with the largest federally qualified health center in the United States, investigators will collect survey data and conduct a randomized experiment on 2,160 individuals (540 families) to evaluate the effectiveness of risk-based messaging and incentives that promote repeated testing for SARS-CoV-2 antibodies. In a 2 x 2 (Messaging x Incentive) factorial experiment, participants complete a comprehensive set of social and behavioral surveys to identify determinants of commitment to testing. Participants are then randomized to receive customized messaging promoting repeated testing. Messaging will focus upon either (1a) household risk or (1b) personal risk of COVID-19. Participants are also randomly assigned to an incentive condition that either (2a) insures against losing baseline rewards for initial testing, or (2b) entry into a lottery with a small chance to win $150 if both tests are completed. Both the loss protection and lottery conditions carry the same incentive costs. Previous work in similar populations demonstrates that adherence to planned health behaviors is higher with insurance-based incentives than cash payments of equal value. This experiment compares insurance-based incentives to lottery incentives that have been shown to be effective in multiple contexts. Finally, the investigators evaluate if social and behavioral determinants of health result in heterogeneous treatment effects that can inform customization of incentive offerings in future programs devoted to increasing uptake of testing or vaccinations among underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children 5 years of age and older

Exclusion Criteria:

* Children under 5 years of age

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2164 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- AltaMed Health, Los Angeles, California, United States

REFERENCES:
- [Derived] Doctor JN, Berg AH, Knight TK, Kadono M, Stewart E, Sonik R, Hochman M, Sood N. Cross-sectional study examining household factors associated with SARS-CoV-2 seropositivity in low-income children in Los Angeles. BMJ Open. 2023 May 31;13(5):e070291. doi: 10.1136/bmjopen-2022-070291. PMID 37258079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2021 and December 2022, potential participants were contacted by phone by a bilingual coordinator and invited to participate in a study about COVID-19.
Pre-assignment Details: We drew a simple random sample of patient households without replacement from AltaMed registry. Each household sampled was contacted to identify eligibility and interest. Households met inclusion criteria if at least one member was a patient at AltaMed and the household contained at least one adult and at least one member 5 to 17 years of age.
Units Other Than Participants: Households
Period: Overall Study
Arm/Group | Personal Risk + Loss Protection | Personal Risk + Lottery Incentive | Family Risk + Loss Protection | Family Risk + Lottery Incentive
Started | 626; 172 Households | 550; 162 Households | 539; 153 Households | 449; 138 Households
Wave 1 Attendance | 308; 85 Households | 285; 82 Households | 286; 78 Households | 203; 62 Households
Wave 2 Attendance | 123; 35 Households | 84; 24 Households | 129; 38 Households | 78; 26 Households
Completed | 123; 35 Households | 84; 24 Households | 129; 38 Households | 78; 26 Households
Not Completed | 503; 137 Households | 466; 138 Households | 410; 115 Households | 371; 112 Households

BASELINE CHARACTERISTICS:
Population: Households who completed baseline survey and agreed to Time 1 antibody testing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Personal Risk + Loss Protection | Personal Risk + Lottery Incentive | Family Risk + Loss Protection | Family Risk + Lottery Incentive | Total
Number analyzed (Participants) | 626 | 550 | 539 | 449 | 2164
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.71 (16.92) | 24.44 (15.64) | 25.58 (16.78) | 26.42 (16.61) | 25.5 (16.51)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 373 | 319 | 307 | 266 | 1265
  Male | 249 | 231 | 231 | 179 | 890
  Non binary | 0 | 0 | 1 | 0 | 1
  Unknown or Not reported | 4 | 0 | 0 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 578 | 501 | 481 | 408 | 1968
  Not Hispanic or Latino | 38 | 46 | 58 | 38 | 180
  Unknown or Not Reported | 10 | 3 | 0 | 3 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 1 | 1 | 6
  Asian | 16 | 14 | 8 | 7 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 5 | 12 | 25 | 18 | 60
  White | 41 | 38 | 39 | 24 | 142
  More than one race | 32 | 16 | 28 | 29 | 105
  Unknown or Not Reported | 528 | 470 | 438 | 369 | 1805
Region of Enrollment [Number; unit: participants]
  United States | 626 | 550 | 539 | 449 | 2164

OUTCOME MEASURES:

1. Primary Outcome: Attendance Rate at Time 2 SARS-CoV-2 Antibody Test
Description: Effectiveness of risk-based messaging and incentives to encourage attendance at Time 2 testing for SARS-CoV-2 antibodies
Time Frame: 6 months
Population: Participants who attended Time 1 antibody testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Personal Risk + Loss Protection | Personal Risk + Lottery Incentive | Family Risk + Loss Protection | Family Risk + Lottery Incentive
Number analyzed (Participants) | 308 | 285 | 286 | 203
Participants | 123 | 84 | 129 | 78
Statistical Analysis 1: Comparison: Personal Risk + Loss Protection vs Personal Risk + Lottery Incentive; Test type: Superiority; p = 0.003, Mixed Models Analysis; Slope = 1.19, 95% CI 2-sided [0.42 to 1.97], Standard Error of Mean 0.40 — Coefficient for mixed effects regression comparing Time 2 attendance to Time 1 attendance for Personal + Loss Protection relative to reference group (Personal + Lottery)
Statistical Analysis 2: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Loss Protection; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 1.46, 95% CI 2-sided [0.68 to 2.24], Standard Error of Mean 0.40 — Coefficient for mixed effects regression comparing Time 2 attendance to Time 1 attendance for Family + Loss Protection relative to reference group (Personal + Lottery)
Statistical Analysis 3: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Lottery Incentive; Test type: Superiority; p = 0.01, Mixed Models Analysis; Slope = 1.11, 95% CI 2-sided [0.26 to 1.96], Standard Error of Mean 0.44 — Coefficient for mixed effects regression comparing Time 2 attendance to Time 1 attendance for Family + Lottery relative to reference group (Personal + Lottery)

2. Secondary Outcome: Social and Behavioral Determinants of Antibody Testing
Description: Characterize barriers to access, bias, risk attitude and incentive preferences assessed through survey responses
Time Frame: 6 months
Population: This analysis was conducted on heads of households who completed the baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Personal Risk + Loss Protection | Personal Risk + Lottery Incentive | Family Risk + Loss Protection | Family Risk + Lottery Incentive
Number analyzed (Participants) | 172 | 162 | 153 | 138
Participants
  Reported the biggest barrier to getting the vaccine is money | 12 | 21 | 17 | 10
  Reported the most trusted source of COVID-19 information is their medical provider | 49 | 47 | 41 | 40
  Scored <=5 on risk aversion scale of 0-10, with 0 being more risk averse and 10 more risk prone | 88 | 75 | 72 | 54
Statistical Analysis 1: Comparison: Personal Risk + Loss Protection vs Personal Risk + Lottery Incentive; Comparison of Time 2 attendance between study arms among respondents who indicated that money was the biggest barrier to getting the vaccine; Test type: Superiority; p = 0.409, Regression, Logistic; Slope = -0.29, 95% CI 2-sided [-0.98 to 0.4], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Loss Protection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.098, Regression, Logistic; Slope = 0.50, 95% CI 2-sided [-0.09 to 1.10], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Lottery Incentive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.982, Regression, Logistic; Slope = 0.01, 95% CI 2-sided [-0.71 to 0.73], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: Personal Risk + Loss Protection vs Personal Risk + Lottery Incentive; Comparison of Time 2 attendance between study arms among respondents who indicated that their medical provider was the most trusted source of COVID-19 information; Test type: Superiority; p = 0.177, Regression, Logistic; Slope = -0.27, 95% CI 2-sided [-0.67 to 0.12], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Loss Protection; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.117, Regression, Logistic; Slope = 0.33, 95% CI 2-sided [-0.08 to 0.74], Standard Error of Mean 0.21
Statistical Analysis 6: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Lottery Incentive; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.809, Regression, Logistic; Slope = 0.05, 95% CI 2-sided [-0.39 to 0.50], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Personal Risk + Loss Protection vs Personal Risk + Lottery Incentive; Comparison of Time 2 attendance between study arms among respondents who scored below or equal to 5 on the risk aversion scale (scale of 0-10, with 0 being more risk averse and 10 being more risk prone); Test type: Superiority; p = 0.847, Regression, Logistic; Slope = 0.04, 95% CI 2-sided [-0.34 to 0.41], Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Loss Protection; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.993, Regression, Logistic; Slope = -0.002, 95% CI 2-sided [-0.39 to 0.38], Standard Error of Mean 0.20
Statistical Analysis 9: Comparison: Personal Risk + Lottery Incentive vs Family Risk + Lottery Incentive; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.671, Regression, Logistic; Slope = -0.09, 95% CI 2-sided [-0.51 to 0.33], Standard Error of Mean 0.22

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Personal Risk + Loss Protection | Personal Risk + Lottery Incentive | Family Risk + Loss Protection | Family Risk + Lottery Incentive
All-Cause Mortality (participants affected / at risk) | 0/626 | 0/550 | 0/539 | 0/449
Serious Adverse Events (participants affected / at risk) | 0/626 | 0/550 | 0/539 | 0/449
Other Adverse Events (participants affected / at risk) | 0/626 | 0/550 | 0/539 | 0/449

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT04901624/Prot_SAP_000.pdf